CLINICAL TRIAL: NCT05348629
Title: Efficacy and Safety of Covid-19 Vaccine in Cardiac Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mina sobhi said fam (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mina sobhi said fam, resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: covid-19 vaccine
Record Dates: First submitted 2022-03-31; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Efficacy and safety of covid-19 vaccine in Cardiac patients

DETAILED DESCRIPTION:
investigate the efficacy and safety of covid-19 vaccine in cardiac patients and its possible assocciated morbidity

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as STEMI undergo PPCI as (Fourth universal definition of myocardial infarction (2018) Kristian Thygesen) 10
* with age range from 18 to 80 years after 1 month of STEMI .

Exclusion Criteria:

* Patients with previous covid infection confirmed by swap or CT chest or ICU addmision.
* Patients with previous covid infection confirmed by qualitative antibdy test .
* Patients with history of anaphylaxis to any component of the vaccine should not take it .
* patients with febrile illness or acute , ongoing infection .
* immunosuppressive diseases .

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ages Eligible for Study : 18 Years to 80 Years Genders Eligible for Study : Male or female
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year
  all cause mortality
Myocardial infarction | one year
  Myocardial infarction
stent thrombosis | one year
  stent thrombosis

SECONDARY OUTCOMES:
Cardiovascular death. Cardiovascular death. Cardiovascular death.Cardiovascular death. cardiovascular death | one year
  Cardiovascular death.
heart failure hospitalization | one year
  heart failure hospitalization
infection by covid-19 | one year
  infection by covid-19
anaphylaxis required hospitalization | one year
  anaphylaxis required hospitalization

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University, Asyut
  - Assiut university, Asyut

IPD SHARING:
Plan to Share IPD: Yes